CLINICAL TRIAL: NCT01508962
Title: PRE-Symptomatic Studies in Amyotrophic Lateral Sclerosis
Acronym: PRESS-ALS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michael Benatar, Professor of Neurology, University of Miami
Other Study IDs: PRESS-ALS
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Disease onset; Disease progression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals (controls)
- Individuals affected with ALS (sporadic or familial)

SUMMARY:
The goal of PRESS-ALS is to study the earliest manifestations of disease in people with early ALS in whom some areas of the body are not yet affected.

ELIGIBILITY:
Inclusion Criteria

ALS group:

* Subject is a male or female, aged at least 18 years.
* Subject is affected with ALS (familial or sporadic).
* Subject has at least one limb in which there is no symptomatic upper and lower motor neuron dysfunction.
* Subject is willing and able to comply with all study procedures.
* Subject agrees to provide signed and dated informed consent form.

Control group:

* Subject is a male or female, aged at least 18 years.
* Subject is not affected with ALS or an ALS-related disorder.
* Subject does not have a family history (i.e., at least 2 biological relatives) of ALS or an ALS-related disorder.
* Subject is willing and able to comply with all study procedures.
* Subject agrees to provide signed and dated informed consent form.

Exclusion Criterion

• Any condition or situation which, in the PI's opinion, could confound the biomarker data or may interfere significantly with the individual's participation and compliance with the study protocol, including but not limited to neurological, psychological and/or medical conditions (e.g., multiple sclerosis, neuropathy, myelopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People affected with ALS (either familial or sporadic) and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Phenoconversion | Every three months over the course of one year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://als-research.org